CLINICAL TRIAL: NCT02023281
Title: The Effects of Exercise on Depression Symptoms Using Levels of Neurotransmitters and EEG as Markers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liberty University (Other)
Collaborators: CommonSpirit Health (Other)
Responsible Party: Principal Investigator, Timothy H. Barclay, Assistant Professor; Licensed Clinical Psychologist, Liberty University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LU4261 from WyndhurstCC; NCT01787201 (obsolete NCT alias)
Record Dates: First submitted 2013-12-23; First posted 2013-12-30 (Estimated); Last update posted 2013-12-30 (Estimated); Status verified 2013-12

CONDITIONS: Depression
Keywords: Depression; Exercise; Neurotransmitters; Catecholimines; EEG
MeSH Terms: conditions — Depression; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): Control group will serve as a wait list and not be exposed to the intervention.
- Experimental Group (Experimental): The experimental group will engage in a mild-moderate level of structured and clinically supervised exercise program for approx. 30-45 mins 2-3 days per week for 12 weeks
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — The experimental group will engage in mild-moderate level of exercise. This program will be structured and clinically supervised. Exercise will take place 2-3 days per week for a duration of 30-45 mins. for 12 weeks.
  Arms: Experimental Group

SUMMARY:
The purpose of this study is to examine the effects of exercise on the symptoms of depression using serum levels of serotonin, catecholamine's, Alpha EEG asymmetry, and self-report of symptoms as markers.

In an attempt to further understand the mechanisms of improved mood through exercise; this study will examine the known factors that contribute to depressed mood in a single study using serotonin and catecholamine levels via blood serum and EEG slow wave asymmetry. Such information can be useful in understanding the overall neurological components of depression and the effects of exercise on the brain in depressed individuals that would make the prescription of exercise a viable treatment option.

DETAILED DESCRIPTION:
There is an increasing demand for clinical effective, safe, and cost conscious forms of treatment for depression. Research shows depression to account for the largest decrease in overall health compared to asthma, angina, arthritis, and diabetes (Maussavi, 2007). The cost of lost productivity at work due to depression is a new focus of research as no current and accurate numbers exist. Stewart, Ricci, Hahn, & Morganstein (2013) were among the first to examine this issue and found that lost productivity due to depression cost an estimated $44 billion dollars per year in spite of current medical treatments commonly prescribed. The lost productivity among those with depression and the low level of treatment suggest that there may be cost effective opportunities for improving depression outcomes within the general workforce and society at large.

The question of value regarding the use of exercise as a treatment for depression has remained a source of investigation in recent years. In cooperation with Centra Health and Liberty University, this study seeks to understand the mechanisms that make exercise a viable treatment in depression by examining self-report of symptoms, serum levels of serotonin and catecholamines (epinephrine, norepinephrin, and dopamine) and frontal slow wave EEG activity as markers. Although these markers have been examined individually in previous studies, this is the only known study that examines each of these components in a single study. Such information can be useful in understanding the overall neurological components of depression and the effects of exercise on the brain in depressed individuals that would make the prescription of exercise a viable treatment in depression.

Multiple trials, meta-analyses, and reviews have been conducted in the attempt to clarify the use of exercise in depressed patients. Research has shown that exercise as a treatment may result in fewer relapses than sertraline (Strohle, 2009). Similar results are indicated when exercise is prescribed as an adjunct treatment with psychotherapy (Balon, Sidhu, & Pankhuree, 2009; Blumenthal, Smith, & Hoffman, 2012; Gill, Womack, & Safranek, 2010). Preliminary characteristics of the ideal dosage of exercise as a treatment have been researched, although a definitive dose-response curve has yet to be produced (Callaghan, Khalil, Morres, & Carter, 2011; Perraton, Kumar, & Machotka, 2010).

Electroencephalographic (EEG) scans have been shown to demonstrate a left frontal bias in alpha (8-12 Hz) and theta (4-7 Hz) wave activity (Allen, Urry, Hitt, & Coan, 2004; Demos, 2005; Iosifescu et al., 2008; Nissen et al., 2006). The up-training or down-training of individual bandwidths in the treatment of depression, anxiety, ADHD, and traumatic brain injury have long been established (La Vaque, 2002). Although there are no established norms for neurotransmitter levels, we know through clinical medication trials that the inhibition of the reuptake of serotonin and or norepinephrine improve mood. Previous studies examining low levels of serotonin and decreased mood have found a correlation between exercise and increased serotonin availability without the use of pharmaceuticals (Chaouloff et al., 1985; Ernst, Olsen, Pinel, Lam, & Christie, 2006; Jacobs & Fornal, 1999). More routine type studies often use neurotransmitter levels as markers (Lande, Williams, Fileta, 2012; Lidberg, Tuck, Asberg, Scalia-Tomba, & Bertilsson, 1985; Mann & Stanley, 1984).

ELIGIBILITY:
Inclusion Criteria:

* primary diagnosis of depression
* 18-65 years of age
* Physically fit to engage in physical exercise

Exclusion Criteria:

* Participants with a history or current symptoms of psychosis
* anticipation of psychiatric medication changes over the course of the study
* Bipolar disorder or other disorder reflecting reality testing impairment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-03; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Scores on the Beck Depression Inventory-II | Pre and post intervention over the 3 month span of the study
  The BDI-II is a 21 item self-report screening tool that measures symptoms of depression.

SECONDARY OUTCOMES:
Serum levels of serotonin and catecholomine | Pre and post intervention over the 3 month span of the study
  Blood collection pre and post intervention for the processing of serum for serotonin and catecholomine.

OTHER OUTCOMES:
Mean EEG alpha frequency data in the pre-frontal cortex. | Pre and post intervention over the 3 month span of the study.
  Participants will have an EEG measuring pre-frontal cortex mean alpha frequency.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy H Barclay, Ph.D., Principal Investigator — Liberty University
Locations (2):
- United States (2):
  - Liberty University, Lynchburg, Virginia
  - Centra Health; Health Works, Lynchburg, Virginia